CLINICAL TRIAL: NCT02987452
Title: Hemodynamic, Autonomic and Inflammatory Answers to Different Types of Exercises in Resistant Hypertensive Patients: an Metabolomic Approach
Brief Title: Acute Effects of Different Exercises on Blood Pressure in Hypertensive Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heitor Moreno Junior (Other)
Responsible Party: Sponsor-Investigator, Heitor Moreno Junior, Full professor, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 55942216.4.0000.5404
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: exercise; resistant hypertension; blood pressure
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- aerobic exercise (Experimental): Aerobic exercise (EA): activity on a treadmill lasting 45 minutes with intensity of 50-60% of maximum heart rate (HR) obtained from ergometer test
  Interventions: Other: aerobic exercise; Other: resistance exercise; Other: combined exercise
- resistance exercise (Active Comparator): resistance exercise (RE): 4 series of 12 repetitions of resistance exercises at moderate intensity (until moderate fatigue), for 45 minutes
  Interventions: Other: aerobic exercise; Other: resistance exercise; Other: combined exercise
- combined exercise (Active Comparator): combined exercise (CE): EA (25 minutes) + ER (20 minutes), with an interval of 2 minutes between sessions totalizing 45 minutes
  Interventions: Other: aerobic exercise; Other: resistance exercise; Other: combined exercise

INTERVENTIONS:
Other: aerobic exercise — Aerobic exercise (EA): activity on a treadmill lasting 45 minutes with intensity of 50-60% of maximum heart rate (HR) obtained from ergometer test
Other: resistance exercise — resistance exercise (RE): 4 series of 12 repetitions of resistance exercises at moderate intensity (until moderate fatigue), for 45 minutes
Other: combined exercise — combined exercise (CE): EA (25 minutes) + ER (20 minutes), with an interval of 2 minutes between sessions totalizing 45 minutes

SUMMARY:
Lifestyle changes might reduce cardiovascular risk due to the decrease in blood pressure (BP). However, whether combining aerobic and resistance exercises affect BP and hemodynamic parameters, as well as arterial stiffness and inflammation markers in resistant hypertensive (RHTN) patients, have not been investigated yet.

DETAILED DESCRIPTION:
Objective: The investigators aim to evaluate the acute effects of aerobic, resistance and combined (aerobic+ resistance) exercise on the BP, hemodynamic and inflammatory parameters, as well as arterial stiffness in RHTN patients compared to mild to moderate hypertensive (HTN) and normotensive (NT) subjects. Design and Methods: This interventional, randomized, single-blind, crossover study will be conducted in 30 patients (RHTN=10, HTN=10, and NT=10) regularly followed in the Outpatient Resistant Hypertension Clinic at UNICAMP- Brazil. All the subjects will be submitted to a previous adaptation of physical activity, especially to determine the load to be implemented in each patient. Then, the modalities of physical exercises (aerobic, resistance and combined) will be randomly performed in three isolated sessions, which will consist of: a) Aerobic exercise (EA): activity on a treadmill lasting 45 minutes with intensity of 50-60% of maximum heart rate (HR) obtained from ergometer test; b) resistance exercise (RE): 4 series of 12 repetitions of resistance exercises at moderate intensity (until moderate fatigue), for 45 minutes; c) combined exercise (CE): EA (25 minutes) + ER (20 minutes), with an interval of 2 minutes between sessions totalizing 45 minutes. Body composition (plethysmography) and cardiorespiratory functional capacity (ergometry) will be determined before the physical training. In addition, the investigators will assess BP recording (by Finometer, office and ambulatory BP), arterial stiffness (by pulse wave velocity, Sphygmocor CPV system), plasma biomarkers (TNF-α, interleukins -1, -6, -10, and -17 by ELISA) in pre and post periods of each physical exercise. Results: Since the physical exercise in its different modalities provides chronic effects on BP in HTN patients, the investigators hypothesized that the isolated (aerobic and resistance) and combined exercise can acutely promote changes in BP levels in RHTN patients when compared to the participants counterparts. Secondarily, some biological mechanisms related to BP control (vascular function and cytokines production) may also be involved in these possible alterations. Conclusion: The investigators expect to define whether a physical exercise program applied to RHTN patients has medical relevance in a realistic clinical setting. These findings may guide the prescription of physical activity as an additional therapeutic approach, in order to decrease the cardiovascular risk associated to these subjects.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis recommended by the AHA Statement on Resistant Hypertension (2008)
* a 6-month period clinic follow-up
* give written informed consent form

Exclusion Criteria:

* secondary Hypertension
* pseudoresistance hypertension (poor medication adherence and white coat hypertension)
* patients with symptomatic ischemic heart disease, impaired renal function, liver disease and history of stroke, myocardial infarction and peripheral vascular diseases, heart failure
* pregnant women
* smoking
* regular physical activity
* mental or physical limitation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure in mmHg | 15 minutes
  systolic blood pressure will be assessed for 15 minutes in baseline, 60 minutes and 24 hours post each interventions.

SECONDARY OUTCOMES:
arterial stiffness | baseline and 60 minutes post each intervention
  by pulse wave velocity, Sphygmocor CPV system
ambulatory blood pressure monitoring | baseline and post each intervention
  ambulatory blood pressure will be assessed in baseline and post each intervention
interleukin 6 | baseline, 60 minutes and 24 hours post each intervention
  interleukin 6 will be assessed by ELISA
interleukin 10 | baseline, 60 minutes and 24 hours post each intervention
  interleukin 10 will be assessed by ELISA
tumor necrosis factor alpha | baseline, 60 minutes and 24 hours post each intervention
  tumor necrosis factor alpha will be assessed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Nayara F. Pires, PhD student, Principal Investigator — University of Campinas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraccari-Pires N, Coelho-Junior HJ, Gambassi BB, Cabral de Faria AP, Ritter AMV, Gasparetti CS, Pioli MR, Ruberti OM, Ferreira-Melo SE, Moreno H, Rodrigues B. Cardiovascular Autonomic Responses to Aerobic, Resistance and Combined Exercises in Resistance Hypertensive Patients. Biomed Res Int. 2022 Apr 20;2022:8202610. doi: 10.1155/2022/8202610. eCollection 2022. PMID 35496038